CLINICAL TRIAL: NCT03254108
Title: A Multicenter, Double-blind, Randomized, Active-controlled, Parallel-group Comparison Clinical Pharmacology Trial to Investigate the Dose of OPC-61815 Injection Equivalent to Tolvaptan 15-mg Tablet in Patients With Congestive Heart Failure
Brief Title: Clinical Pharmacology Trial to Investigate the Dose of OPC-61815 Injection Equivalent to Tolvaptan 15-mg Tablet in Patients With Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 263-102-00001; JapicCTI-173676 (Other: Japic)
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- OPC-61815 injection 2mg (Experimental): Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 2 mg.
  Interventions: Drug: OPC-61815 injection 2mg
- OPC-61815 injection 4mg (Experimental): Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 4 mg.
  Interventions: Drug: OPC-61815 injection 4mg
- OPC-61815 injection 8mg (Experimental): Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 8 mg.
  Interventions: Drug: OPC-61815 injection 8mg
- OPC-61815 injection 16mg (Experimental): Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 16 mg.
  Interventions: Drug: OPC-61815 injection 16mg
- Tolvaptan tablet 15mg (Active Comparator): Once daily for 5 days tolvaptan 15-mg tablet will be orally administered, followed immediately by 1-hour intravenous administration of placebo.
  Interventions: Drug: Tolvaptan tablet 15mg

INTERVENTIONS:
Drug: OPC-61815 injection 2mg — Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 2 mg.
  Arms: OPC-61815 injection 2mg
Drug: OPC-61815 injection 4mg — Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 4 mg.
  Arms: OPC-61815 injection 4mg
Drug: OPC-61815 injection 8mg — Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 8 mg.
  Arms: OPC-61815 injection 8mg
Drug: OPC-61815 injection 16mg — Once daily for 5 days placebo tablet will be orally administered, followed immediately by intravenous administration of OPC-61815 at 16 mg.
  Arms: OPC-61815 injection 16mg
Drug: Tolvaptan tablet 15mg — Once daily for 5 days tolvaptan 15-mg tablet will be orally administered, followed immediately by 1-hour intravenous administration of placebo.
  Arms: Tolvaptan tablet 15mg

SUMMARY:
The dose for intravenous administration of OPC-61815 achieving tolvaptan exposure equivalent to that for oral administration of tolvaptan 15-mg tablet will be investigated by administering OPC-61815 injection 2 to 16mg or tolvaptan 15-mg oral tablet to subjects with congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are currently on treatment with any of the following diuretics

   * Loop diuretics equivalent to furosemide tablet or fine granules at a dose of 40 mg/day or higher
   * Concomitant use of a loop diuretic and a thiazide diuretic (including thiazide analogs) at any dose
   * Concomitant use of a loop diuretic and an aldosterone antagonist or potassium-sparing diuretic agent at any dose
2. Subjects with congestive heart failure in whom lower limb edema, pulmonary congestion, and/or jugular venous distension due to volume overload is present
3. Subjects who are currently hospitalized or who are able to be hospitalized during the trial

Exclusion Criteria:

1. Subjects with acute heart failure
2. Subjects with a history of hypersensitivity to any of ingredients of OPC-61815 or tolvaptan
3. Subjects who are unable to sense thirst or who have difficulty with fluid intake

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kanto, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 74 subjects were screened for this trial, 13 were screen failures, and 61 were randomly assigned to one of the treatment groups. One subject assigned to the OPC-61815 16-mg group was withdrawn due to dehydration before initiation of the trial drug administration; therefore, 60 subjects received at least 1 dosing of the trial drug.
Period: Overall Study
Arm/Group | OPC-61815 Injection 2mg | OPC-61815 Injection 4mg | OPC-61815 Injection 8mg | OPC-61815 Injection 16mg | Tolvaptan Tablet 15mg
Started | 13 | 12 | 12 | 12 | 12
Received Treatment | 13 | 12 | 12 | 11 | 12
Completed | 13 | 10 | 12 | 11 | 9
Not Completed | 0 | 2 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 1
Not completed — AST/ALT is increased to 3 times upper limit of normal or higher | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all subjects treated with the investigational medicinal product (IMP) at least once
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-61815 Injection 2mg | OPC-61815 Injection 4mg | OPC-61815 Injection 8mg | OPC-61815 Injection 16mg | Tolvaptan Tablet 15mg | Total
Number analyzed (Participants) | 13 | 12 | 12 | 11 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (9.5) | 74.5 (11.9) | 72.2 (9.9) | 77.9 (3.8) | 74.8 (8.9) | 74.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 3 | 2 | 19
  Male | 8 | 8 | 7 | 8 | 10 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 12 | 12 | 11 | 12 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 13 | 12 | 12 | 11 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of OPC-41061 on Day 1
Time Frame: Baseline, 1, 1.5, 2, 4, 6, 12 24 hours after the start of administration of investigational drug
Population: Subjects treated with the IMP at least once and had at least 1 data of primary endpoint after IMP administration
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OPC-61815 Injection 2mg | OPC-61815 Injection 4mg | OPC-61815 Injection 8mg | OPC-61815 Injection 16mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 12
ng/mL | 41.4 (11.4) | 98.6 (43.7) | 149 (61.7) | 282 (96.0) | 325 (194)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC24h) on Day 1
Time Frame: Baseline, 1, 1.5, 2, 4, 6, 12 24 hours after the start of administration of investigational drug
Population: Subjects treated with the IMP at least once and had at least 1 data of primary endpoint after IMP administration
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OPC-61815 Injection 2mg | OPC-61815 Injection 4mg | OPC-61815 Injection 8mg | OPC-61815 Injection 16mg | Tolvaptan Tablet 15mg
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 12
ng*h/mL | 356 (157) | 983 (563) | 1340 (522) | 2400 (1030) | 2850 (1580)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the start of IMP administration up to 15 days
Description: Subjects who received at least 1 dose of IMP were included in the safety analysis.
Arm/Group | OPC-61815 Injection 2mg | OPC-61815 Injection 4mg | OPC-61815 Injection 8mg | OPC-61815 Injection 16mg | Tolvaptan Tablet 15mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12 | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 7/13 | 7/12 | 4/12 | 8/11 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 Injection 2mg (N=13) | OPC-61815 Injection 4mg (N=12) | OPC-61815 Injection 8mg (N=12) | OPC-61815 Injection 16mg (N=11) | Tolvaptan Tablet 15mg (N=12)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 Injection 2mg (N=13) | OPC-61815 Injection 4mg (N=12) | OPC-61815 Injection 8mg (N=12) | OPC-61815 Injection 16mg (N=11) | Tolvaptan Tablet 15mg (N=12)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 1 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 2 | 0 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Jugular vein distension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT03254108/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT03254108/SAP_001.pdf